CLINICAL TRIAL: NCT06568263
Title: Celiac Disease and Quality of Life in Children and Adolescents (CeliaQLife)
Acronym: CeliaQLife
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Janne Anita Kvammen, PhD, Principal Investigator, Oslo University Hospital
Other Study IDs: 591377
Record Dates: First submitted 2024-08-12; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Celiac Disease in Children; Nutritional Deficiency; Quality of Life
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood, urine and feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Celiac disease: Children diagnosed with celiac disease on a gluten-free diet
- Healthy: Healthy children on a regular diet

SUMMARY:
Celiac disease is a disorder commonly diagnosed during childhood. The treatment is a lifelong gluten-free diet. Both the condition and the diet can influence the children's physical and emotional well-being.

The main goal of this observational study is to learn about nutritional status in a group of children with celiac disease compared to a group of healthy children.

The nutritional assessment includes information on diet, biochemical measurement, and body composition. Quality of life will also be assessed.

The study can contribute to ensure good health and well-being in children on a gluten-free diet.

DETAILED DESCRIPTION:
* A 24-hour dietary recall will be done by a clinical dietician to assess intake of energy and micro- and macronutrients.
* Blood will be drawn for assessment of vitamin- and mineral status.
* Feces and urine samples will be collected to measure gluten immunogenic peptides (GIP) to assess exposure to gluten.
* A self-developed interview will be used for assessment of adherence to the gluten-free diet and compared with the results from a 11-item questionnaire.
* Weight and height will be measured.
* Bone mineral density and body composition will be measured by dual-energy x-ray absorptiometry (DXA).
* Health-related quality of life (QOL) will be measured by the PedsQL.

ELIGIBILITY:
Inclusion Criteria:

* eating a regular diet

Exclusion Criteria:

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Age: 6-18 years
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Iron deficiency will be assessed from hemoglobin and ferritin in children with celiac disease and in healthy children. Differences in the prevalences of iron deficiency between children with celiac disease and healthy children will be described. | All participants will be assessed once. The study time frame is from August 2024 until December 2025.
  Blood samples will be analyzed for blood hemoglobin and serum ferritin.

CONTACTS AND LOCATIONS:
Overall Officials: Janne A Kvammen, Phd, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo
  - University of Oslo, Oslo

IPD SHARING:
Plan to Share IPD: Undecided